CLINICAL TRIAL: NCT01350635
Title: Evaluation of BM32, a Recombinant Hypoallergenic Grass Pollen Vaccine, by Skin Testing
Brief Title: Skin Test Study of BM32
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biomay AG (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS-BM32-001
Record Dates: First submitted 2011-05-07; First posted 2011-05-10 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Hypersensitivity
Keywords: Specific Immunotherapy; Grass pollen vaccine; Allergy; Grass Pollen Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: BM32 — BM32 will be applied in sterile phosphate buffer solution. Drug will be applied in concentrations of 11,33 and 100 micrograms/ml

SUMMARY:
The aim of the present skin test study CS-BM32-001 is to evaluate whether the BM32 proteins exhibit low/no allergenic activity when applied by skin prick- and atopy patch testing to grass pollen allergic patients

DETAILED DESCRIPTION:
BM32 is a hypoallergenic grass pollen allergy vaccine which consists of an aluminum hydroxide-adsorbed equimolar mix of four active ingredients, BM321, BM322, BM325 and BM326. The four active ingredients are purified recombinant proteins containing non-allergenic peptides from the four major timothy grass pollen allergens, Phl p 1 (BM321), Phl p 2 (BM322), Phl p 5 (BM325) and Phl p 6 (BM326) which are fused to the PreS domain of hepatitis B virus, a protein used in childhood vaccines. BM32 holds promise not to induce IgE mediated immediate type (e.g. anaphylactic reactions) or T-cell mediated late phase side effects during immunotherapy.

The aim of the present skin test study CS-BM32-001 is to evaluate whether the BM32 proteins due to their low/absent IgE- and T cell-reactivity exhibit low/no allergenic activity when applied by skin prick- and atopy patch testing to grass pollen allergic patients (n=60). This study will therefore provide important information for immunotherapy studies based on BM32.

ELIGIBILITY:
Inclusion Criteria:

* Positive history of grass pollen allergy and positive skin prick test reaction to grass pollen extract
* Age between 18 and 60 years
* Subjects must have a standard health care insurance
* Subject must appear capable to understand and comply with all relevant aspects of the study protocol

Exclusion Criteria:

* pregnancy or breast feeding
* autoimmune diseases, immune defects including immuno- suppression, immune-complex-induced immunopathies
* contra-indication for adrenaline
* severe general maladies, malignant diseases
* patients under long-term treatment with systemic corticosteroids, immunosuppressive drugs, tranquilizers or psychoactive drugs
* contra-indications for skin prick testing such as: skin inflammation in the test area, urticaria facticia, unstable or uncontrolled bronchial asthma (30)
* use of beta-blockers
* participation in another clinical trial within one month prior to the study; however, participation during the previous month solely in the form of blood donation without other interventions will be acceptable
* risk of non-compliance with the study procedure and restrictions
* use of oral H1 antihistamines within the previous 3 days, oral Ketotifen within the previous 5 days and topical corticosteroids in the test area within the previous 14 days.
* systemic (short-term) corticosteroids within the previous 14 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
wheal size of immediate type skin reactions to the mix of BM32 proteins wheal size of immediate type skin reactions to the wheal size of immediate type skin reaction to the mix of BM32 proteins | 20 minutes
  For skin prick testing a drop of the test solution will be placed on the subjects´ skin at a distance of at least 2 cm between individual application points. The skin will be pricked with sterile prick lancets. Reactions will be recorded after 20 minutes by measuring the diameters of the wheal. Wheals of more than 3 mm diameter will be regarded as positive reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University, Vienna, Vienna, Austria